CLINICAL TRIAL: NCT00811434
Title: Improvement of Cognitive Function and Healthcare -Related Quality of Life After Lactulose Treatment in Children With Chronic Liver Disease
Brief Title: Study of Lactulose in Children With Chronic Liver Disease
Acronym: MHE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: funding period ended
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 0808-19; Clarian Grant VFR-279
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Minimal Hepatic Encephalopathy
Keywords: encephalopathy; pediatric liver disease; pediatric cirrhosis; serum ammonia levels
MeSH Terms: conditions — Brain Diseases | interventions — Lactulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactulose (Active Comparator): 3 months of Lactulose therapy based on pt. weight
  Interventions: Drug: Lactulose
- placebo (Placebo Comparator): 1.5 ml/kg day po of sugar water placebo for three months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Lactulose — 1.5cc/kg/day po for three months
  Arms: Lactulose
Drug: placebo — 1.5 ml sugar water/kg day for three months
  Arms: placebo

SUMMARY:
Pediatric patients with chronic liver disease may have Minimal Hepatic Encephalopathy(MHE)which can cause changes in behavior,intelligence and neurological function.By utilizing cognitive and developmental testing we will determine if patients have MHE. If so, we will trial 3 months of blinded placebo or Lactulose treatment followed by a washout period with no treatment. At this time patients are re-tested and then begin another three month period switching to the opposite treatment of first 3 months.Final cognitive/developmental testing will determine if Lactulose treatment has any effect on MHE.

DETAILED DESCRIPTION:
In addition ,serum ammonia levels will be obtained at beginning of study,post-washout and at end of study to evaluate Lactulose effect on serum ammonia.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MHE as result of cognitive, developmental testing, pediatric pt. with cirrhosis as evidenced by imaging/biopsy

Exclusion Criteria:

* patients with neurological,psychiatric or unstable medical conditions which may contribute to impaired cognitive function.
* patients with known hearing or vision difficulties.
* those patients who do not speak English will be excluded.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Girish Subbarao, M.D., Principal Investigator — Indiana University
Locations (1):
- James Whitcomb Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Informed consent was obtained on the first subject 1/16/2009 and recruitment continued until study closure in November 2010.
Pre-assignment Details: Two subjects were withdrawn prior to randomization.Two did not meet entry criteria.
Groups:
- Lactulose First, Then Placebo: Lactulose therapy based on weight; Washout; placebo therapy of 1.5ml/kg/day
- Placebo First, Then Lactulose: Placebo therapy of 1.5ml/kg/day; washout; lactulose therapy based on weight
Period: First Intervention
Arm/Group | Lactulose First, Then Placebo | Placebo First, Then Lactulose
Started | 7 | 5
Completed | 4 | 5
Not Completed | 3 | 0
Period: Washout (1 Month)
Arm/Group | Lactulose First, Then Placebo | Placebo First, Then Lactulose
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Lactulose First, Then Placebo | Placebo First, Then Lactulose
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: all aprticipants who were randomized to receive treatment
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Minimal Hepatic Encephalopathy (MHE) in Children With Cirrhosis
Description: failure of one cognitive function test indicates presence of MHE
Time Frame: baseline
Measure: Number; unit: participant
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 12
participant | 6

2. Secondary Outcome: Health Related Quality of Life (HRQOL)
Description: HRQOL administered to parents prior to treatment
Time Frame: baseline
Population: data not collected as planned
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 0

3. Secondary Outcome: Effeccts of Lactulose Treatment on MHE as Measaured by Cognitive Function
Description: MHE as measured by failure of one or more cognitive test
Time Frame: before and after each treatment period
Population: data not collected as planned
Arm/Group | Lactulose | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Total of 23 months
Description: Assessed at both in person patient visits and phone call follow up
Arm/Group | Lactulose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes